CLINICAL TRIAL: NCT03267368
Title: Pilot Trial of Clinical Implementation of a Comprehensive Care Program for Early Stage Medically Inoperable/Borderline Operable Lung Cancer Patients Undergoing Stereotactic Radiotherapy (SBRT)
Brief Title: Comprehensive Care Program SBRT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment. 1 pt. enrolled & withdrew at 6 wk follow-up. No further enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Inga Grills, Professor, Residency Program Director, Chief Thoracic Section, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-151
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer; Smoking; Copd
Keywords: Comprehensive Care Program; Stereotactic Radiotherapy
MeSH Terms: conditions — Lung Neoplasms; Smoking; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, intervention, outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive Care Program (Experimental): Pulmonary rehab and smoking cessation program/intervention/assessment
  Interventions: Behavioral: Comprehensive Care Program

INTERVENTIONS:
Behavioral: Comprehensive Care Program — Pulmonary rehabilitation and smoking cessation

SUMMARY:
Pulmonary (lung) rehabilitation, which is done under the guidance of lung specialists/therapists. It includes breathing exercises, physical exercises, and exercises to increase tolerance of activity (stamina). This type of lung rehab has been shown to improve symptoms, quality of life, breathing, and walking distance. It has also been shown to decrease hospitalization and death rates in chronic obstructive pulmonary disease (COPD) and lung cancer patients.

Comprehensive Care Management Program (CCMP), a program that includes educational sessions for tobacco cessation, phone calls, and a home action plan has also demonstrated benefit in addition to the pulmonary rehabilitation.

In this study, the investigators have an opportunity to identify and intervene with COPD patients. The vast majority of early stage lung cancer patients are much more scared of their cancer than their COPD. Upon identification of COPD and recognition of patient tobacco habits for patients planned to undergo SBRT, interventions can potentially be made that will reduce COPD hospitalization rates, second primary lung cancer rates, and likely death rates. The interventions are broadly available and relatively easily instituted and include the following: seeing a doctor to diagnose their other underlying illness or illnesses (both respiratory and cardiovascular), smoking cessation if they are smokers, and CCMP's and pulmonary rehabilitation which have shown measurable COPD benefits in prior trials.

DETAILED DESCRIPTION:
Primary objective: To evaluate the technical feasibility and delivery of a comprehensive program that leads to prevention and management of symptoms of COPD in early stage lung cancer patients undergoing curative therapy, promotes and leads to smoking cessation, and evaluates potentially unknown cardiopulmonary co-morbid or therapeutically-induced diseases in the cancer patient.

Secondary objective(s):

1. To document overall survival of patients undergoing lung SBRT plus preventative care, including evaluation and treatment by a pulmonologist and cardiologist in combination with a tobacco cessation program (for those currently smoking or within 6 months of quitting), and pulmonary rehabilitation. Overall survival and other tumor recurrence and survival endpoints will be compared to historical controls.
2. To evaluate quality of life (QOL) changes of patients undergoing lung SBRT with usual care plus evaluation and treatment by a pulmonologist and cardiologist in combination with a tobacco cessation program (for those currently smoking), and pulmonary rehabilitation.
3. To evaluate primary tumor control, regional control, distant metastasis and progression-free and cause-specific survival rates.
4. To evaluate toxicity rates, including pulmonary and cardiotoxicity after SBRT. Diagnosis and management of cardiopulmonary toxicities may be greater for these patients undergoing routine evaluation by specialist physicians.
5. To evaluate smoking cessation rates after employing an Ask, Assist and Refer method for smoking cessation.
6. To evaluate second primary lung cancer rates and compare them to historical controls.
7. To evaluate changes in pulmonary function, 6-minute walk test and V02 max values with participation in pulmonary rehabilitation.
8. To document hospitalization rates after SBRT using these preventative care strategies.
9. To explore the impact of SBRT on ventilation and changes in functional lung using 4-Dimensional computed tomography(4DCT) before and after SBRT.
10. To study the potential impact of SBRT on cardiac function using pre-and post-SBRT EKG and echocardiography.

Patients for this study will be identified in the Radiation Oncology department as being planned to receive SBRT for their lung cancer. All eligibility will be reviewed. Once a patient is deemed eligible and reviewed and signed the informed consent, he/she will be asked to complete the smoking questionnaire available on the state of Michigan (MI) Quitline. If a patient is deemed eligible and decline to enroll, they will be asked to voluntarily complete the American Heart Association (AHA) Smoking Quiz as an eligible patient exit form. Following their completion of this quiz, they will be asked again if they are certain of their desire to decline the study. All enrolled patients will also complete the AHA smoking quiz.

Before Treatment:

All eligibility will be confirmed and pre-treatment standard staging activities (history and physical, zubrod, weight, thoracic surgeon evaluation, chest CT with contrast, 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT), Pulmonary Function Test, bloodwork and pregnancy safety evaluation) will have occurred.

A baseline pulmonologist referral will be made within 4 weeks before/after SBRT.

A baseline cardiologist referral will be made within 4 weeks before/after SBRT.

Baseline EKG and echocardiogram (ECHO) will be done prior to the 1st fraction of SBRT.

Pulmonary rehab baseline assessment including a 6 Minute Walk Test, oxygen consumption (VO2 max) will occur prior to treatment.

Charlson Comorbidity Index Evaluation will occur prior to treatment.

Quality of life, Depression, Anxiety, and Craving Assessment questionnaires will be completed.

Subject will also have a urine or saliva Nicotine evaluation and enrollment in the Michigan Tobacco Quitline program which requires a cell phone or tablet owned by the patient. This is a free service within Michigan, available to any smokers, not specific for the study.

SBRT will take place as prescribed by the treating radiation oncologist within the standard parameters. On-Treatment Visits (OTV) will occur weekly during the SBRT and include a history and physical, zubrod (performance score), weight, hospitalization and smoking assessment, and urine or saliva Nicotine evaluation . As part of the study, nicotine replacement is required to be ordered as is daily visits/calls with a smoking cessation specialist.

After completion of radiotherapy, the subject will have weekly visits/calls with the smoking cessation specialist for 6 weeks.

Post-Treatment visits:

At 6 weeks post SBRT-the patient will come back to the radiation oncology clinic for a history and physical, zubrod, and weight. The patient also have pulmonary function testing (PFT), adverse event reporting, 6 minute walk test and pulmonary rehab per plan developed pre-treatment, hospitalization and smoking assessment #1 Research 4DCT, not diagnostic, will be obtained at this visit and done in the radiation oncology department.

The following testing will happen, as stated at 3, 6, 9, 12, 18, 24, and then annually per standard. Procedures specific to this study will be completed at 24 months. Any annual testing is standard and that data will be used at the time of analysis so it is captured in the patient consent and table of events.

* History and physical exam (3, 6, 9, 12 months)
* Performance status and weight (6, 9, 12, 18, 24, + annual)
* Cardiologist evaluation with EKG/ECHO (6 months)
* CT chest with contrast (3, 6, 9, 12, 18, 24, 30, 36, 42, 48 months, then annual)
* FDG PET (3 months)
* PFT (3, 6, 12, 18, 24 months, then annual)
* Bloodwork- Complete blood count (CBC)/Chemistries (3 months)
* Tumor evaluation (3, 6, 9, 12, 18, 24, then annual)
* Adverse event (side effects) evaluation (3, 6, 9, 12, 18, 24, and annual)
* 2nd primary lung cancer documentation (not patient test-study specific notation)-(12, 24 months then annual)
* 6-minute walk test, V02 Max (3, 6, 12, 24, + annual)
* QOL Assessment (3, 6, 9, 12, 18, 24, + annual)
* Hospitalization and Smoking Assessment (3, 6, 9, 12, 18, then every 6 months to 36 months then annual)
* Urine/Saliva Nicotine evaluation (6, 12, 24 months, then annual if needed)
* Depression, Anxiety, and Craving Assessments (6, 12 months) •# 2 Research 4DCT (6 months)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of non-small cell lung cancer (NSCLC), including the following types: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, large cell neuroendocrine carcinoma, NSCLC not otherwise specified (NOS) *Patients with large cell neuroendocrine tumors must have staging MRI of the brain (or CT with IV contrast if MRI contraindicated) due to the high rate of central nervous system (CNS) metastasis
* American Joint Committee on Cancer (AJCC) Lung 7th Edition clinical Stage T1-T2 N0 M0 with tumor less than or equal to 5 cm size
* Patient will undergo lung SBRT with curative intent
* Zubrod 0 - 2
* Patient evaluated by a Thoracic surgeon and deemed medically inoperable or borderline operable (candidate for only limited lung resection, either wedge resection or segmentectomy) within 8 weeks. For borderline operable patients, patient has seen both thoracic surgery and radiation oncology and has declined surgical intervention
* Baseline pulmonary function tests confirm that patient would medically qualify for Pulmonary Rehabilitation based on current guidelines. This means patient either has COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) II-IV or meets the non-COPD qualifying definition below (FVC, forced expiratory volume at one second (FEV1), or diffusing capacity of lung for carbon monoxide (DLCO) < 65%) AND/OR patient is a current smoker (a non-COPD patient that is a smoker still has a modifiable risk factor; this will be a rare condition).
* Patient is at least 18 years of age
* Patient is a non-pregnant female and/or a female or male practicing adequate means of birth control
* Patient has either peripheral or central lung tumor location that is radiographically identifiable, with central locations as defined by either Radiation Therapy Oncology Group (RTOG) 0236 or RTOG 0813 criteria and will be likely to meet dose volume constraints for central mediastinal structures using one of the allowable dose fractionation schedule.

Exclusion Criteria:

* Patient has had a synchronous primary malignancy, including lung cancer within 2 years, excluding non-invasive cancers or early stage skin cancers
* Patient has had prior lung or thoracic radiotherapy, including prior lung SBRT
* Patient is planned to receive adjuvant systemic therapy for the management of this lung malignancy
* Does not own a functional mobile/cellular communication device (cellular phone, iPhone or iPad), or is not willing to incur any potential plan-specific additional charges
* Patients who cannot perform the prescribed rehabilitation and assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementation of Comprehensive Care program | 6 months after enrollment
  % of enrolled patients who complete study visits

SECONDARY OUTCOMES:
Overall Survival | an average of 10 years
  Time from diagnosis to recurrence or death
Smoking Cessation | 6 months after enrollment
  % of participants who quit smoking

CONTACTS AND LOCATIONS:
Overall Officials: Inga Grills, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Beaumont Health System, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No